CLINICAL TRIAL: NCT01092260
Title: Glomerular Filtration Rate in Children - a Methodological Study With Iohexol Clearance
Brief Title: Renal Function Measurements in Children
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/741
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Renal Function Disorder
Keywords: Glomerular Filtration Rate; Kidney disease; Child; Iohexol; Cystatin C; Measurement of kidney function in children
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum and urine

SUMMARY:
The purpose of this study is to validate a feasible, safe and reliable iohexol plasma clearance method in routine monitoring of the renal function (GFR) in children.

Different parameters of renal function will be compared to the gold standard multiple sample points procedure of iohexol clearance.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years
* Clinical indication for measurement of glomerular filtration rate

Exclusion Criteria:

* Previous serious reaction on Iohexol

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with clinical indication for measurement of renal function
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Tondel, MD, Principal Investigator — Haukeland University Hospital, Bergen, Norway
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Salvador CL, Flemmen PTK, Tondel C, Bliksrud YT, Tsui EFF, Brun A, Bjerre A, Morkrid L. Renal function, sex and age influence purines and pyrimidines in urine and could lead to diagnostic misinterpretation. Mol Genet Metab. 2023 Nov;140(3):107649. doi: 10.1016/j.ymgme.2023.107649. Epub 2023 Jul 5. PMID 37517327
- [Derived] Eide TT, Hufthammer KO, Brun A, Brackman D, Svarstad E, Tondel C. Accuracy of single intravenous access iohexol GFR in children is hampered by marker contamination. Sci Rep. 2021 Dec 1;11(1):23224. doi: 10.1038/s41598-021-02759-1. PMID 34853376
- [Derived] Salvador CL, Tondel C, Rowe AD, Bjerre A, Brun A, Brackman D, Bolstad N, Morkrid L. Renal Function Influences Diagnostic Markers in Serum and Urine: A Study of Guanidinoacetate, Creatine, Human Epididymis Protein 4, and Neutrophil Gelatinase-Associated Lipocalin in Children. J Appl Lab Med. 2017 Nov 1;2(3):297-308. doi: 10.1373/jalm.2016.022145. PMID 33636843
- [Derived] Salvador CL, Tondel C, Rowe AD, Bjerre A, Brun A, Brackman D, Morkrid L. Estimating glomerular filtration rate in children: evaluation of creatinine- and cystatin C-based equations. Pediatr Nephrol. 2019 Feb;34(2):301-311. doi: 10.1007/s00467-018-4067-3. Epub 2018 Aug 31. PMID 30171354
- [Derived] Tondel C, Salvador CL, Hufthammer KO, Bolann B, Brackman D, Bjerre A, Svarstad E, Brun A. Iohexol plasma clearance in children: validation of multiple formulas and single-point sampling times. Pediatr Nephrol. 2018 Apr;33(4):683-696. doi: 10.1007/s00467-017-3841-y. Epub 2017 Nov 13. PMID 29134449
- [Derived] Tondel C, Bolann B, Salvador CL, Brackman D, Bjerre A, Svarstad E, Brun A. Iohexol plasma clearance in children: validation of multiple formulas and two-point sampling times. Pediatr Nephrol. 2017 Feb;32(2):311-320. doi: 10.1007/s00467-016-3436-z. Epub 2016 Jul 1. PMID 27369694